CLINICAL TRIAL: NCT04879394
Title: Pain Sensitivity and Psychological Profile of Chronic Low Back Pain Patients: Implications for a Personalized Treatment Approach
Brief Title: Pain Sensitivity and Psychological Profile of Chronic Low Back Pain Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Minho (Other)
Collaborators: Hospital de Braga (Other); Clinical Academic Center (2CA-Braga) (Other)
Responsible Party: Principal Investigator, Patrícia Ribeiro Pinto, Researcher, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2CA2019
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis (Experimental): 4 weekly hypnosis sessions, aiming at pain control and distress management. The 90 min. sessions will be conducted in group format by a doctorate-level psychologist trained in hypnosis. Contents will be detailed on hypnosis protocols to ensure standardization.
  Interventions: Other: Hypnosis
- Control (No Intervention): Receives standard care as usual. Assessments will be made in the same time points as experimental group, but without undergoing intervention.

INTERVENTIONS:
Other: Hypnosis — 4 weekly hypnosis sessions, aiming at pain control and distress management. The 90 min. sessions will be conducted in group format by a doctorate-level psychologist trained in hypnosis. Contents will be detailed on hypnosis protocols to ensure standardization.
  Arms: Hypnosis

SUMMARY:
This study aims to characterize pain sensitivity and psychological profile of CLBP patients in comparison with pain free adults, and explore their predictive role on hypnosis outcomes, an effective intervention for pain control.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a very prevalent condition, associated with high disability and financial costs. Pain sensitization and psychological status have been associated with symptom severity and treatment outcomes, but their prognostic value is not yet well established.

This is a Prospective Randomized Controlled Trial, with an experimental (hypnosis) and one control group (standard care), and 5 assessment points: baseline, post intervention, 1, 3 and 6 months follow-up. Participants will be 160 CLBP patients and 50 pain free adults, assessed on sociodemographic, clinical, pain, disability, psychophysical (Quantitative Sensory Testing) and psychological variables.

This work will contribute to a better knowledge of the mechanisms underlying CLBP and of the patient characteristics that can predict treatment outcomes after hypnosis. The findings have the potential to improve patient-targeted treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* persistent or recurrent low back pain lasting over 3 months

Exclusion Criteria:

* pain due to other causes (e.g. fibromyalgia, fracture)
* back surgery in the previous 6 months or planned in the following 6 months
* debilitating organic, psychiatric or neurological conditions (e.g. cancer, schizophrenia, dementia)
* disability compensation or litigation related to CLBP
* unavailability to commit to the hypnosis sessions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity at 1 week as assessed by Numeric Rating Scale (NRS) | 1 week post-intervention
  Pain intensity assessed by NRS
Pain intensity at 1 month as assessed by NRS | 1 month post-intervention
  Pain intensity assessed by NRS
Pain intensity at 3 months as assessed by NRS | 3 months post-intervention
  Pain intensity assessed by NRS
Pain intensity at 6 months as assessed by NRS | 6 months post-intervention
  Pain intensity assessed by NRS

SECONDARY OUTCOMES:
Pain interference at 1 week as assessed by the Brief Pain Inventory (BPI) | 1 week post-intervention
  Pain interference assessed by the BPI
Pain interference at 1 month as assessed by the BPI | 1 month post-intervention
  Pain interference assessed by the BPI
Pain interference at 3 months as assessed by the BPI | 3 months post-intervention
  Pain interference assessed by the BPI
Pain interference at 6 months as assessed by the BPI | 6 months post-intervention
  Pain interference assessed by the BPI
Functionality at 1 week as assessed by the Oswestry Low Back Pain Disability Questionnaire (ODI) | 1 week post-intervention
  Functionality assessed by the ODI
Functionality at 1 month as assessed by the ODI | 1 month post-intervention
  Functionality as assessed by the ODI
Functionality at 3 months as assessed by the ODI | 3 months post-intervention
  Functionality assessed by the ODI
Functionality at 6 months as assessed by the ODI | 6 months post-intervention
  Functionality assessed by the ODI
Quality of life at 1 week as assessed by the EuroQol Quality of Life Questionnaire (EQ-5D-5L) | 1 week post-intervention
  Quality of life assessed by the EQ-5D-5L
Quality of life at 1 month as assessed by the EQ-5D-5L | 1 month post-intervention
  Quality of life assessed by the EQ-5D-5L
Quality of life at 3 months as assessed by the EQ-5D-5L | 3 months post-intervention
  Quality of life assessed by the EQ-5D-5L
Quality of life at 6 months as assessed by the EQ-5D-5L | 6 months post-intervention
  Quality of life assessed by the EQ-5D-5L
Emotional distress at 1 week as assessed by the Hospital Anxiety and Depression Scale (HADS) | 1 week post-intervention
  Emotional distress assessed by HADS
Emotional distress at 1 month as assessed by the Hospital Anxiety and Depression Scale (HADS) | 1 month post-intervention
  Emotional distress assessed by HADS
Emotional distress at 3 months as assessed by the Hospital Anxiety and Depression Scale (HADS) | 3 months post-intervention
  Emotional distress assessed by HADS
Emotional distress at 6 months as assessed by the Hospital Anxiety and Depression Scale (HADS) | 6 months post-intervention
  Emotional distress assessed by HADS
Optimism at 1 week as assessed by the Life Orientation Test (LOT) | 1 week post-intervention
  Optimism assessed by LOT
Optimism at 1 month as assessed by LOT | 1 month post-intervention
  Optimism assessed by LOT
Optimism at 3 months as assessed by LOT | 3 months post-intervention
  Optimism assessed by LOT
Optimism at 6 months as assessed by LOT | 6 months post-intervention
  Optimism assessed by LOT
Pain catastrophizing at 1 week as assessed by the Pain Catastrophizing Scale (PCS) | 1 week post-intervention
  Pain catastrophizing assessed by PCS
Pain catastrophizing at 1 month as assessed by PCS | 1 month post-intervention
  Pain catastrophizing assessed by PCS
Pain catastrophizing at 3 months as assessed by PCS | 3 months post-intervention
  Pain catastrophizing assessed by PCS
Pain catastrophizing at 6 months as assessed by PCS | 6 months post-intervention
  Pain catastrophizing assessed by PCS

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia R Pinto, PhD, Principal Investigator — University of Minho
Locations (1):
- Hospital de Braga, Braga, Portugal